CLINICAL TRIAL: NCT07163741
Title: Validity and Reliability of the 6-Minute Pegboard and Ring Test in Patients With Coronary Artery Disease
Status: Not yet recruiting | Type: Observational
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Meral Boşnak Güçlü, Prof. Dr., Gazi University
Other Study IDs: 2025-1418
Record Dates: First submitted 2025-09-02; First posted 2025-09-09 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Coronary Artery Disease (CAD)
Keywords: coronary artery disease; 6 minute pegboard and ring test; functional upper extremity exercise capacity
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient with coronary artery disease group: The maximal exercise capacity for the upper limb will be evaluate by CPET and performed on the arm ergometer in addition to the upper limb functional exercise capacity will be evaluate by 6 minute pegboard and ring test.

SUMMARY:
Coronary artery disease, a cardiovascular disease, causes significant mortality and morbidity. Due to the impairment of arterial blood flow in coronary artery disease, the heart muscle cannot receive an adequate blood supply during exercise, resulting in symptoms such as chest pain, shortness of breath, and fatigue, which can lead to a decrease in exercise capacity. The 6-Minute Pegboard and Ring Test is a simple, rapid, and inexpensive assessment tool used to evaluate upper extremity exercise capacity. The purpose of this study was to assess the validity and reliability of the 6-Minute Pegboard and Ring Test in patients with coronary artery disease.

DETAILED DESCRIPTION:
Coronary artery disease, a cardiovascular disease, causes significant mortality and morbidity. Due to the impairment of arterial blood flow in coronary artery disease, the heart muscle cannot receive an adequate blood supply during exercise, resulting in symptoms such as chest pain, shortness of breath, and fatigue, which can lead to a decrease in exercise capacity. The 6-Minute Pegboard and Ring Test is a simple, rapid, and inexpensive assessment tool used to evaluate upper extremity exercise capacity. The purpose of this study was to assess the validity and reliability of the 6-Minute Pegboard and Ring Test in patients with coronary artery disease.

Within the scope of the study, at least 32 patients diagnosed with coronary artery disease (CAD) will undergo the "6-Minute Pegboard and Ring Test" (6-PBRT), which assesses upper extremity functional exercise capacity, and the upper extremity cardiopulmonary exercise test, which assesses maximal exercise capacity, on two separate days, 48 hours apart. The 6-Minute Pegboard and Ring Test will be repeated twice, 1 hour apart, by the same evaluator. Before and after the test, heart rate (HR), oxygen saturation, respiratory frequency, arm fatigue, general fatigue, and dyspnea parameters will be assessed. In the 6-PBRT, heart rate and oxygen saturation will be measured with a pulse oximeter (Soulfix Fingertip Oximeter Pulse Oxygen Meter, ABD); fatigue and dyspnea will be assessed with the Modified Borg Scale (MBS); and respiratory frequency will be assessed by counting the number of breaths taken per minute. Patients' respiratory muscle strength will be assessed using a portable oral pressure monitor (Micro Medical MicroRM, UK); respiratory function tests will be performed using a spirometer (Cosmed, Class II/Internally Powered Equipment, Italy); and peripheral muscle strength will be assessed using a portable handheld dynamometer (JTECH Power Track Commander, Baltimore, USA). Patients' quality of life will be assessed using the "Heart Quality of Life Scale in Coronary Artery Disease Patients." All assessments and tests will be explained in detail to the patient beforehand.

ELIGIBILITY:
Inclusion Criteria:

* Individuals diagnosed with coronary artery disease by conventional angiography or computed tomography coronary angiography,

  * Clinically stable,
  * Ages between 18 and 85,
  * Volunteering to participate in the study will be included in the study.

Exclusion Criteria:

* Individuals diagnosed with heart failure,

  * Those diagnosed with moderate-to-severe valvular disease,
  * Those with a history of orthopedic, neurological, or pulmonary disease that could affect exercise testing and exercise capacity,
  * Those with contraindications to exercise testing according to the American College of Sports Medicine (ACSM) criteria,
  * Those with a history of coronary artery bypass surgery will not be included in the study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 32 patients diagnosed with coronary artery disease will be recruited.
Sampling Method: Probability Sample
Enrollment: 32 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2026-06-06 (Estimated); Study Completion 2026-09-25 (Estimated)

PRIMARY OUTCOMES:
Upper Limb Functional Exercise Capacity | Through study completion, an average of 1 year
  The 6-minute pegboard ring test will be performed using two wooden blocks, each set at shoulder level and 20 cm above, for a total of 20 rings. Before the test, participants are instructed to simultaneously place wooden rings from the lower blocks onto the upper blocks using both hands and to continue the same process in reverse for 6 minutes. The goal of the test is to move as many rings as possible from bottom to top and top to bottom within six minutes. The total number of rings is recorded. Participants receive standard verbal encouragement each minute. Heart rate, blood pressure, shortness of breath, upper extremity fatigue, and overall fatigue are measured before and immediately after the test.
Maximal Exercise Capacity | Through study completion, an average of 1 year
  Maximal Exercise capacity will be evaluated with Cardiopulmonary Exercise testing. The Cardiopulmonary Exercise Testing will be applied according to American Thoracic Society (ATS) and European Respiratory Society (ERS) criteria.

SECONDARY OUTCOMES:
Respiratory Muscle Strength Assessment | Through study completion, an average of 1 year
  To assess respiratory muscle strength, voluntary maximal inspiratory pressure (MIP) and maximal expiratory pressure (MEP) will be measured using an electronic, portable oral pressure measuring device (Micro Medical MicroRM, UK) according to ATS/ERS criteria. Participants will be seated upright in a chair and asked to inhale deeply to their total lung capacity, then exhale rapidly and forcefully to their residual lung volume. To measure MEP, patients will be asked to exhale to their residual lung capacity, then inhale rapidly and forcefully to their total lung capacity. During the measurement, participants will be given verbal prompts to support the measurement. Measurements will continue until the difference between each best measurement is less than 5% or 5% H₂O. The participant's best measurement will be recorded. As a result of the measurements, the equations prepared by Evans and his colleagues will be used to calculate the expected values appropriate to the age and gender of the
Respiratory Function Assessment | Through study completion, an average of 1 year
  Dynamic lung volumes will be assessed using a spirometer (Cosmed, Class II/Internally Powered Equipment, Italy) in an upright sitting position with the nose closed, according to the criteria of the American Thoracic Society (ATS) and the European Respiratory Society (ERS). Pulmonary function testing will measure FVC, FEV1, FEV1/FVC, peak expiratory flow (PEF), and FEF 25-75% flow rate. The best of three technically acceptable maneuvers with 95% agreement will be selected for statistical analysis.
Peripheral Muscle Strength Assessment | Through study completion, an average of 1 year
  Patients' peripheral muscle strength will be assessed using a portable handheld dynamometer (JTECH Power Track Commander, Baltimore, USA) for the upper extremities (deltoid muscle strength) and quadriceps muscle strength for the lower extremities (quadriceps muscle strength). Patients will be seated unsupported, with the arm in 90-degree abduction and flexion, and quadriceps muscle strength will be assessed with the knee in 90-degree extension. These measurements will be repeated three times on the right and left sides, and the best measurements will be recorded in Newtons (N) and used in the analysis. The reference equations of Andrews et al. will be used to calculate expected values based on age, gender, and body weight.
Assessment of Shortness of Breath and Fatigue | Through study completion, an average of 1 year
  Patients' perception of shortness of breath and fatigue at rest and during activities of daily living will be assessed using the modified Borg Scale. Additionally, shortness of breath and general body and arm fatigue during exercise testing will be assessed using the modified Borg Scale.
Assessment of Chronotropic Response | Through study completion, an average of 1 year
  A chronotropic response is the increase in heart rate in response to physical activity or exercise. Conversely, the absence of an increase in heart rate due to exercise or an inadequate increase in heart rate is defined as chronotropic insufficiency [14]. Chronotropic insufficiency can be assessed using the chronotropic index, which uses the maximal heart rate achieved during exercise testing and the resting heart rate.
Heart Quality of Life (HeartQoL) Scale | Through study completion, an average of 1 year
  The scale consists of 14 items and two subscales: physical (10 items) and emotional (4 items). Each item on the HeartQoL Scale is scored between 0 and 3, with 3 indicating "no discomfort" and 0 indicating "very much discomfort."

CONTACTS AND LOCATIONS:
Overall Officials: Aslınur ÇAKIR, MSc., Study Chair — Gazi University; Naciye Sevim, Pt., Principal Investigator — Gazi University; Meral Boşnak Güçlü, Prof. Dr., Study Director — Gazi University
Locations (1):
- Gazi University Faculty of Health Sciences Department of Cardiopulmonary Physiotherapy and Rehabilitation, Ankara, Çankaya 06490, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Miller MR, Crapo R, Hankinson J, Brusasco V, Burgos F, Casaburi R, Coates A, Enright P, van der Grinten CP, Gustafsson P, Jensen R, Johnson DC, MacIntyre N, McKay R, Navajas D, Pedersen OF, Pellegrino R, Viegi G, Wanger J; ATS/ERS Task Force. General considerations for lung function testing. Eur Respir J. 2005 Jul;26(1):153-61. doi: 10.1183/09031936.05.00034505. No abstract available. PMID 15994402
- [Background] Evans JA, Whitelaw WA. The assessment of maximal respiratory mouth pressures in adults. Respir Care. 2009 Oct;54(10):1348-59. PMID 19796415
- [Background] Nashef SA, Roques F, Sharples LD, Nilsson J, Smith C, Goldstone AR, Lockowandt U. EuroSCORE II. Eur J Cardiothorac Surg. 2012 Apr;41(4):734-44; discussion 744-5. doi: 10.1093/ejcts/ezs043. Epub 2012 Feb 29. PMID 22378855